CLINICAL TRIAL: NCT04220983
Title: PRAGMA (Prostate Radio Ablation Guided by Magnetic Resonance Imaging Acquisition) in Metastatic Prostate Cancer
Acronym: PRAGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-04020263
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MR-Guided Prostate SBRT (Other)
  Interventions: Radiation: MR-Guided Prostate SBRT

INTERVENTIONS:
Radiation: MR-Guided Prostate SBRT — Prostate SBRT has become a standard of care for the treatment of localized prostate cancer. Radiation is delivered to the prostate and seminal vesicles in 5 treatment sessions (fractions). Doses ranging from 35-45 Gy in 5 fractions have demonstrated good outcomes with acceptable toxicity when planning is delivered appropriately.

SUMMARY:
Patients with metastatic prostate cancer can undergo MRI-guided prostate Stereotactic body radiation therapy (SBRT) without significant adverse events, similar to what has been reported for patients with localized prostate cancer. We hypothesize that prostate SBRT will be well-tolerated in metastatic prostate cancer patients, with quality of life outcomes similar to what has been reported in non-metastatic prostate cancer patients.

DETAILED DESCRIPTION:
The MRidian ViewRay offers delivery of prostate SBRT with real-time MR guidance, which provides superior soft-tissue differentiation with excellent visualization of the prostate. This ViewRay platform offers the ideal setting for this study, that aims at precisely delivering prostate SBRT with a simultaneous integrated boost (when indicated) to visible nodules.

In this study, we hope to demonstrate the safety and feasibility of using 36.25 Gy in 5 fractions, plus a simultaneous integrated boost (when indicated), in patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of prostate adenocarcinoma
* Age ≥ 18
* Must have biopsy-proven metastatic prostate cancer

Exclusion Criteria:

* History of prior pelvic radiation (external beam or brachytherapy)
* Inability to undergo MRI
* AUA score >20
* For patients on systemic therapy, enrollment must be within six months of start of therapy unless exception is made by protocol PIs.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MR-Guided Prostate SBRT
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MR-Guided Prostate SBRT
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Subjects With Adverse Events Will be Collected
Description: Treatment will be deemed safe if there is no more than 3 acute Grade 3 gasterointestinal/genitourinary events within the first 30 days after treatment completion. Adverse events can be unexpected or expected, related to treatment.
Time Frame: baseline, 3-6months and at 9-12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | MR-Guided Prostate SBRT
Number analyzed (Participants) | 22
Participants
  Baseline | 22
  3-6 months | 18
  9-12 months | 17

2. Secondary Outcome: Change in Quality of Life Questionnaires Will be Assessed.
Description: Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. There are 5 domains, urinary incontinence, urinary Irritative/Obstructive, Bowel, Sexual function and Hormonal. For each domain, the scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes. QOL assessments will occur at baseline, 3-6 months, and at 9-12 months.
Time Frame: baseline, 3-6months and at 9-12 months.
Population: 1 patient was not assessed at baseline time point, as the patient had a foley, 4 patients were not assessed at 3-6 months time point, 5 patients were not assessed at 9-12 months time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MR-Guided Prostate SBRT
Number analyzed (Participants) | 22
score on a scale
  Baseline : Urinary incontinence: number analyzed (Participants) | 21
  Baseline : Urinary incontinence | 80.6 (22.1)
  Baseline : Urinary Irritative/Obstructive: number analyzed (Participants) | 21
  Baseline : Urinary Irritative/Obstructive | 83.4 (15.5)
  Baseline : Bowel: number analyzed (Participants) | 21
  Baseline : Bowel | 96.8 (5.5)
  Baseline : Sexual Function: number analyzed (Participants) | 21
  Baseline : Sexual Function | 8.6 (14.1)
  Baseline : Hormonal: number analyzed (Participants) | 21
  Baseline : Hormonal | 74.1 (19.3)
  3-6 months : Urinary incontinence: number analyzed (Participants) | 18
  3-6 months : Urinary incontinence | 84.75 (2.93)
  3-6 months : Urinary Irritative/Obstructive: number analyzed (Participants) | 18
  3-6 months : Urinary Irritative/Obstructive | 84.55 (0.47)
  3-6 months : Bowel: number analyzed (Participants) | 18
  3-6 months : Bowel | 92.2 (3.2)
  3-6 months : Sexual Function: number analyzed (Participants) | 18
  3-6 months : Sexual Function | 4.7 (2.8)
  3-6 months : Hormonal: number analyzed (Participants) | 18
  3-6 months : Hormonal | 62.7 (8.05)
  9-12 months : Urinary incontinence: number analyzed (Participants) | 17
  9-12 months : Urinary incontinence | 84.9 (3.08)
  9-12 months : Urinary Irritative/Obstructive: number analyzed (Participants) | 17
  9-12 months : Urinary Irritative/Obstructive | 82.8 (0.75)
  9-12 months : Bowel: number analyzed (Participants) | 17
  9-12 months : Bowel | 91.6 (3.68)
  9-12 months : Sexual Function: number analyzed (Participants) | 17
  9-12 months : Sexual Function | 5.7 (2.05)
  9-12 months : Hormonal: number analyzed (Participants) | 17
  9-12 months : Hormonal | 72.8 (0.95)

3. Secondary Outcome: Change in The International Prostate Symptom Score (I-PSS) Will be Assessed.
Description: The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicatingincreasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
Time Frame: baseline, 3-6months and at 9-12 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MR-Guided Prostate SBRT
Number analyzed (Participants) | 22
score on a scale
  Baseline | 10.7 (7.9)
  3-6 months: number analyzed (Participants) | 18
  3-6 months | 9 (1.2)
  9-12 months: number analyzed (Participants) | 17
  9-12 months | 12.2 (1.12)

ADVERSE EVENTS:
Time Frame: Baseline, 3-6 months, 9-12 months
Arm/Group | MR-Guided Prostate SBRT
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MR-Guided Prostate SBRT (N=22)
Diffused Pruritic Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MR-Guided Prostate SBRT (N=22)
Fatigue (General disorders) | 12 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (22)
Bladder incontinence (Renal and urinary disorders) | 4 (22)
Constipation (Gastrointestinal disorders) | 2 (22)
Hot flashes (Vascular disorders) | 9 (22)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (22)
Weak Urine Stream (Renal and urinary disorders) | 2 (22)
Nocturia (Renal and urinary disorders) | 2 (22)
Urinary Frequency (Renal and urinary disorders) | 15 (22)
Appetite change (Gastrointestinal disorders) | 1 (22)
Anxiety (Nervous system disorders) | 1 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04220983/Prot_SAP_000.pdf